CLINICAL TRIAL: NCT07313267
Title: Effectiveness of an Intervention Programme Using Alternative Sports for the Recovery of Motor Learning and the Improvement of Physical and Mental Health in Primary School Students.
Brief Title: Intervention With Alternative Sports for Physical and Mental Improvement in Primary School Children
Acronym: Renew
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, María P. Pezoa Fuentes, Doctor of Physical Activity Sciences, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UCM-IN-25214; UCM-IN-25214 (Other Grant/Funding Number: UNIVERSIDAD CATÓLICA DEL MAULE, CHILE.)
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Primary School Students; Healthy
Keywords: physical fitness; motor skills; children; physical interventions; alternative sports
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The trial is designed as a cluster-randomized trial with randomization units: course groups. The minimum clinically relevant difference in body fat percentage has been defined as 3 percentage points (Δ = 3), with an estimated standard deviation of 5. A significance level of α = 0.05 (two-tailed) and statistical power of 80% were assumed. An average cluster size of n = 35 students and a loss/adherence rate of 15% were considered. Based on recent literature on CRTs in school children, an intracluster correlation coefficient (ICC) = 0.03 was assumed.
  With these assumptions, ≈ 44 students per arm are needed in an individual trial. Adjusting for cluster effect with ICC = 0.03, the size per arm increases to ≈ 88 students. Then, considering 15% losses, the final size per arm is ≈ 104 students. To cover this with average group sizes of 35, 3 courses/clusters per arm (6 clusters in total) will be needed, implying 210 enrolled students (105 intervention / 105 control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with alternative sports (Experimental): The experimental group will hold 90-minute sessions twice a week for two months. Each two-week block will be dedicated to an alternative sport (flag football, ultimate frisbee, korfball, and kin-ball).
  Interventions: Other: Intervention with Alternative Sports (kin-ball, korfball, ultimate frisbee and flag football))
- Control Group, traditional classes. (Active Comparator): The control group (CG) will only participate in the initial and final evaluations, continuing with their traditional physical education classes without modifications, distributed in two weekly sessions of 90 minutes each.
  The classes incorporate sports and motor activities that involve collaborative sports and games.
  Interventions: Other: Intervention with regular classes from the school curriculum

INTERVENTIONS:
Other: Intervention with Alternative Sports (kin-ball, korfball, ultimate frisbee and flag football)) — The RENUÉVATE intervention will be implemented by previously trained physical education teachers. It will last for two months, with sessions held twice a week. The sessions will take place during the school day, in physical education classes, and will last 90 minutes. Each two-week block will be dedicated to an alternative team sport (flag football, ultimate frisbee, korfball, and kin-ball). The physical load for each session is as follows:
  Warm-up (15 min): general mobility and specific exercises to prepare for the sport in question, maintaining an intensity of 50-60% HRmax; RPE 9-11.
  Main part (65 min): practice of the alternative sport through games and technical/tactical progressions. An intensity of 65-80% HRmax will be prescribed; RPE 12-15, with active breaks between tasks.
  Cool down (10 min): relaxation, stretching, and group reflection activities with a light intensity <50% HRmax; RPE ≤ 9.
  Arms: Intervention with alternative sports
Other: Intervention with regular classes from the school curriculum — The intervention will be implemented by physical education teachers who have been trained in the project's objectives, methodology, and values. The training will include a standardized manual and a two-hour weekly practical session to ensure fidelity in the program's implementation. In addition, weekly monitoring meetings will be held with the research team to resolve questions and ensure consistency across schools.
  Arms: Control Group, traditional classes.

SUMMARY:
The objective of this clinical trial is to determine whether a school-based intervention involving alternative sports can improve physical fitness, motor skills, and psychological well-being in elementary school students. The main question to be answered is:

Can participating in a physical intervention involving alternative sports help children improve their strength, speed, endurance, motor skills, and enjoyment of physical activity? For 8 weeks, during physical education classes, researchers will compare an intervention with alternative sports (korfball, flag football, kin-ball, and ultimate frisbee) with the usual classes that students receive according to their study program, to see if alternative sports improve physical and psychological aspects.

Participants must:

* Perform physical and motor tests to determine their initial physical condition
* Complete a questionnaire to determine their level of enjoyment during physical activity.
* Actively participate in an 8-week intervention during physical education classes.
* Monitor their level of physical activity during classes using a device (accelerometer).
* Authorize the use of their first semester grades.
* At the end of the intervention, physical and motor tests will be performed again to assess progress and physical changes.

For eight weeks, researchers will conduct a study in physical education classes to compare two types of teaching: one based on alternative sports (such as korfball, flag football, kin-ball, and ultimate frisbee) and another with traditional school program classes to see if children improve physically and psychologically.

DETAILED DESCRIPTION:
The RENUEVATE study is a randomized controlled cluster trial with a parallel group design and repeated measurements, developed using a quantitative approach. The study follows the CONSORT guidelines for randomized cluster trials and has been approved by the Scientific Ethics Committee of the Catholic University of Maule, Chile (Resolution No. 112/2025). All procedures comply with the principles of the Declaration of Helsinki.

Randomization is performed at the educational establishment level in order to reduce the risk of contamination between participants. Three urban establishments in the city of Talca, Chile, representative of different administrative and socioeconomic contexts (municipal and privately subsidized), are randomly assigned to the intervention group (IG) or control group (CG). In each establishment, one sixth-grade class is assigned to the IG and another to the CG, making a total of six clusters.

Participants in the intervention group receive the RENUEVATE program, a school physical activity intervention integrated into regular physical education classes. The program is implemented during the academic period by previously trained physical education teachers, using a standardized manual that ensures the fidelity of the intervention. Teachers receive initial training and periodic supervision from the research team.

The intervention is based on the use of alternative sports (flag football, ultimate frisbee, korfball, and kin-ball), selected for their ability to promote moderate to vigorous physical activity, motor skill development, cooperation, inclusion, and gender equality. Each session follows a standardized structure that includes warm-up, main development, and cool-down phases, prescribing the intensity necessary to achieve adequate levels of physical effort during the central phase. The fidelity and dose of the intervention are monitored through session records, subjective perception of effort, and heart rate monitoring in a subsample of participants.

The control group continues with the regular physical education curriculum taught by the school, without modifications or exposure to the intervention content, participating only in pre- and post-intervention assessments.

Assessments are conducted at two points in time: before the start of the intervention (baseline) and at the end of the program, during the school day and by previously trained assessors, ideally blinded to group assignment. Primary and secondary outcomes include variables of physical fitness, motor skills, physical activity levels, body composition, enjoyment of physical activity, and health-related quality of life, assessed using validated instruments widely used in children. A detailed description of the variables and measurement instruments is presented in the corresponding sections of the registry.

The sample size was estimated to detect a clinically relevant difference in the percentage of body fat between groups, considering the cluster design and an expected intraclass correlation. Statistical analysis will be performed under the intention-to-treat principle, using mixed-effects models that allow for the hierarchical structure of the data and repeated measurements over time, adjusting for baseline values and relevant covariates. The procedures for handling missing data and sensitivity analyses are predefined in the study protocol.

ELIGIBILITY:
The inclusion criteria for participants are as follows:

* Be enrolled in the assigned school.
* Have no motor problems that prevent participation in the physical activities proposed for the development of alternative sports.
* Have completed ≥ 85% of the sessions. The exclusion criteria
* Not having taken the initial or final tests.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Motor competence | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  It will be assessed using the Motorishe Basiskompetenzen (MOBAK) battery, which evaluates body control (balance, rolling, jumping) and object control (throwing, catching, bouncing, dribbling), used in schoolchildren aged 10 to 12.
  For throwing and catching tasks, children have 6 attempts (no trial attempts), in which the number of successes, i.e., successful attempts, is recorded. These are then scored: 0 to 2 successes, 0 points; 3 to 4 successes, 1 point; and 5 to 6 successes, 2 points.
  -For the tasks of driving with the hand, driving with the foot, balancing, rolling, jumping, and running. Children have 2 attempts to complete the task (no trial attempts). The scoring of these tests is based on a dichotomous scale (0 = not achieved, 1 = achieved), in which the number of successful attempts is recorded (never achieved = 0 points; achieved once = 1 point; achieved twice = 2 points).
  The score from 0 to 8 determines the level of basic motor skills in a differentiated manner.
Physical fitness | A measurement will be taken at the start of the intervention on day 1 (pre-test) and another assessment will be carried out at the end of the intervention on day 16 (post-test).
  Physical fitness will be assessed, using tests that have been widely validated in school populations: For cardiorespiratory capacity, a 6-minute walk test will be used to estimate VO₂max; Lower limb muscle strength will be assessed using the squat jump (SJ) and counter-movement jump (CMJ) on a force platform, and handgrip strength will be assessed using a Camry EH101 hydraulic dynamometer, recognized for its high reliability.
Enjoyment | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  Enjoyment of physical activity was assessed using the Spanish version of the Physical Activity Enjoyment Scale (PACES). This scale consists of 16 items. Responses were collected on a 5-point Likert scale (1 = Strongly disagree to 5 = Strongly agree). The score is obtained by calculating the average of the 16 items.
  The total score ranges from 16 to 80, with higher values indicating greater enjoyment.

SECONDARY OUTCOMES:
Body Composition (Bioelectrical Impedance Analysis) | It will be evaluated on day 1 (pre-test) and day 16 (post-test)
  Name of the measure: Body fat percentage Description: Body composition will be assessed using eight-electrode tetrapolar bioelectrical impedance analysis with the InBody 570® device. The outcome corresponds to body fat percentage obtained according to the manufacturer's standardized measurement protocol.
  Unit of measure: Percentage (%) Range: 0 to 100 percent. Direction of outcome: Lower values indicate a better outcome.
Morphological variables (Body Height) | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  Name of the measure: Body height Description: Body height measured following ISAK standardized protocols by an ISAK Level II anthropometrist.
  Unit of measure: Meters (m) Range: No predefined minimum or maximum values. Direction of outcome: Not applicable (descriptive anthropometric measure).
Morphological variables (Body Weight) | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  Name of the measure: Body weight Description: Body weight measured according to the International Society for the Advancement of Kinanthropometry (ISAK) standardized protocols by an ISAK Level II anthropometrist.
  Unit of measure: Kilograms (kg) Range: No predefined minimum or maximum values. Direction of outcome: Not applicable (descriptive anthropometric measure).
Morphological variables (Body Mass Index) | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  Name of the measure: Body Mass Index Description: Body Mass Index calculated as body weight in kilograms divided by height in meters squared (kg/m²), using measurements obtained according to ISAK standardized protocols by an ISAK Level II anthropometrist.
  Unit of measure: Kilograms per square meter (kg/m²) Range: No predefined minimum or maximum values. Direction of outcome: Lower values indicate a more favorable body composition.
Morphological variables (Waist Circumference) | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  Name of the measure: Waist circumference Description: Waist circumference measured according to ISAK standardized protocols by an ISAK Level II anthropometrist.
  Unit of measure: Centimeters (cm) Range: No predefined minimum or maximum values. Direction of outcome: Lower values indicate a more favorable central adiposity profile.
Physical activity level (objective) | It will be evaluated on day 1 (pre-test) and day 16 (post-test)
  Name of the measure: Moderate-to-vigorous physical activity Description: Physical activity level will be objectively assessed using ActiGraph wGT3X-BT triaxial accelerometers. Data will be processed using ActiLife software and the GGIR package in R. Time spent in moderate-to-vigorous physical activity will be calculated using validated pediatric cut-off points. The outcome corresponds to the average daily minutes of moderate-to-vigorous physical activity.
  Unit of measure: Minutes per day (min/day) Range: 0 to no predefined maximum value. Direction of outcome: Higher values indicate a better outcome (higher physical activity level).
Level of physical activity (self-reported) | It will be measured on day 1 (pre-test) and day 16 (post-test).
  This will be assessed using the Physical Activity Questionnaire for Adolescents (PAQ-A).
  Description of the scale:
  The Physical Activity Questionnaire for Adolescents is a self-administered instrument designed to assess the overall level of physical activity of adolescents during the previous seven days, including physical activity performed at school, during leisure time, and on weekends.
  Scale range:
  The total score ranges from 1 to 5 and is calculated as the average score of the questionnaire items.
  Interpretation of scores:
  Higher scores indicate a higher level of physical activity. Lower scores indicate a lower level of physical activity.
Health-related quality of life | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  Name of the scale: KIDSCREEN-27 Health-Related Quality of Life Questionnaire Scale description:The KIDSCREEN-27 Health-Related Quality of Life Questionnaire is a self-administered instrument designed to assess health-related quality of life in children and adolescents. It evaluates five dimensions: Physical Well-being, Psychological Well-being, Autonomy and Parent Relations, Social Support and Peers, and School Environment.
  Scale range: Each dimension is scored on a 5-point Likert scale, and dimension scores are transformed into standardized values ranging from 0 to 100.
  Interpretation of scores: Higher scores indicate better health-related quality of life. Lower scores indicate poorer health-related quality of life.
  Direction of outcome: Higher scores represent a better outcome.

OTHER OUTCOMES:
Sociodemographic Characteristics (Covariates) | It will be evaluated on day 1 (pre-test) and day 16 (post-test).
  Name of the measure: Family socioeconomic status Description: Family socioeconomic status will be assessed using a questionnaire completed by parents or legal guardians. The questionnaire will collect information on parental educational level, household income, and family structure. These variables will be combined to classify participants into predefined socioeconomic status categories for descriptive and adjustment purposes.
  Unit of measure: Categorical variable (low, medium, high socioeconomic status). Range: Not applicable. Direction of outcome: Not applicable (descriptive covariate)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio N Merellano Navarro, Doctor, Study Director — Universidad Católica del Maule
Locations (1):
- Universidad Católica del Maule, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
Yes, inpatient data will be shared, specifically the data supporting the results of the publication. Study participants will be assigned a code, and that data will be shared.
Supporting Information: Study Protocol
Time Frame: Individual patient data will be available from July 2026 to December 2026.
Access Criteria: * The criteria that must be met for data to be shared.
  * The study design must be experimental, using a controlled trial.
  * The intervention group must be between 10 and 12 years old.
  * Statistical methods will be analyzed using mixed linear models, considering the fixed effect of the group (GI vs. GC), baseline, age, and sex, and including a random effect by school cluster to adjust for intraclass correlation.
  * The mechanism for sharing data is to submit a written request by email, indicating the reasons for the data request, providing a summary of the project, and disclosing the statistical analysis to be performed.
  * Once the document has been reviewed and approved by the principal investigator, a data exchange agreement will be signed.

REFERENCES:
- [Result] Zurita-Ortega, F., Ubago-Jiménez, J. L., Ibáñez, E. M., González-Valero, G., & Alonso Vargas, J. M. Effects of a physical education programme based on kin ball on body mass index and basic physical skills in students with down syndrome. (2025). https://doi.org/10.12800/ccd.v20i63.2211
- [Result] Vaquero-Solís, M., Tapia-Serrano, M. A., Moreno-Díaz, M. I., Cerro-Herrero, D., & Sánchez-Miguel, P. A. Exploratory analysis of physical activity in self-objectification and body image of adolescents. Cultura, Ciencia y Deporte, (2021). 16(48), 199-206. https://doi.org/10.12800/CCD.V16I48.1724
- [Result] Stewart, A., Marfell-Jones, M., Olds, T., & de Ridder, J. International Standards for Anthropometric Assessment. (2011). ISAK.
- [Result] Muñoz Troncoso, F., Becerra Peña, S., & Riquelme, E. Elaboración y validación psicométrica del cuestionario de convivencia escolar para la no violencia (CENVI). Estudios Pedagógicos (Valdivia), (2017). 43(3), 205-223. https://doi.org/10.4067/S0718-07052017000300012
- [Result] Moya-Mata, I., Ruiz-Sanchis, L., Martín-Ruiz, J., & Ros-Ros, C. Physical activity represented in physical education textbooks for elementary education. Movimento, (2019). 25(1). https://doi.org/10.22456/1982-8918.89296
- [Result] Morales-Campo PT, Perez-Munoz S, Lopez-Garcia S, Diez-Fernandez P, Rodriguez-Cayetano A. New alternative proposal in physical education: Touchtennis as a racket sport in schools. Front Sports Act Living. 2025 Mar 3;7:1545994. doi: 10.3389/fspor.2025.1545994. eCollection 2025. PMID 40098917
- [Result] Migueles, J. H., Rowlands, A. V., Huber, F., Sabia, S., & Van Hees, V. T. GGIR: A Research Community-Driven Open Source R Package for Generating Physical Activity and Sleep Outcomes From Multi-Day Raw Accelerometer Data. Journal for the Measurement of Physical Behaviour, 2019. 2(3), 188-196. https://doi.org/10.1123/jmpb.2018-0063
- [Result] Martins S, Augusto C, Martins MRO, Jose Silva M, Okan O, Dadaczynski K, Duarte A, Fronteira I, Ramos N, Rosario R. Adaptation and validation of the Digital Health Literacy Instrument for Portuguese university students. Health Promot J Austr. 2022 Oct;33 Suppl 1:390-398. doi: 10.1002/hpja.580. Epub 2022 Feb 17. PMID 35124876
- [Result] Markovic J, Bubanj S, Sekeljic G, Pavlovic S, Radenkovic M, Stankovic D, Petkovic E, Aksovic N, Radenkovic O, Preljevic A, Bjelica B, Petrovic V, Sinanovic S, Tomovic M. Efficiency of an Alternative Physical Education Program for the Lower Grades of Elementary School Children. Children (Basel). 2023 Oct 6;10(10):1657. doi: 10.3390/children10101657. PMID 37892320
- [Result] Marfell-Jones, M. J., Stewart, A., & de Ridder, J. H. International standards for anthropometric assessment. (2012). International Society for the Advancement of Kinanthropometry.
- [Result] Leuschner M, Grauduszus M, Friesen D, Ferrari N, Klaudius M, Joisten C. The 6-minute Run Test: Validation and Reference Equations for Adults. Int J Sports Med. 2024 Mar;45(3):222-230. doi: 10.1055/a-2206-5291. Epub 2023 Dec 19. PMID 38113901
- [Result] Lettink A, Altenburg TM, Arts J, van Hees VT, Chinapaw MJM. Systematic review of accelerometer-based methods for 24-h physical behavior assessment in young children (0-5 years old). Int J Behav Nutr Phys Act. 2022 Sep 8;19(1):116. doi: 10.1186/s12966-022-01296-y. PMID 36076221
- [Result] Herrmann, C. MOBAK 1-4. Test zur Erfassung Motorischer Basiskompetenzen für die Klassen 1-4 (2018). Hogrefe.
- [Result] Chen C, Weyland S, Fritsch J, Woll A, Niessner C, Burchartz A, Schmidt SCE, Jekauc D. A Short Version of the Physical Activity Enjoyment Scale: Development and Psychometric Properties. Int J Environ Res Public Health. 2021 Oct 20;18(21):11035. doi: 10.3390/ijerph182111035. PMID 34769552
- [Result] Budler LC, Pajnkihar M, Ravens-Sieberer U, Barr O, Stiglic G. The KIDSCREEN-27 scale: translation and validation study of the Slovenian version. Health Qual Life Outcomes. 2022 Apr 21;20(1):67. doi: 10.1186/s12955-022-01973-3. PMID 35448993